CLINICAL TRIAL: NCT01496352
Title: A Randomized, Double-blind, Placebo Controlled, Safety, Tolerability, and Pharmacokinetic Dose Escalation Study of DFA-02 in Patients Undergoing Colorectal Surgery
Brief Title: DFA-02 in Patients Undergoing Colorectal Surgery
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Collaborators: Duke Clinical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DFA-02-CD-002
Record Dates: First submitted 2011-12-15; First posted 2011-12-21 (Estimated); Results first posted 2014-09-01 (Estimated); Last update posted 2014-09-01 (Estimated); Status verified 2014-08

CONDITIONS: Surgical Site Infection
Keywords: Surgical site infection; Colorectal surgery
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DFA-02 (Experimental): Progressive cohorts of 10 subjects (8 active, 2 placebo) receiving 10, 20 , 30 or 40 mL of DFA-02 or matching placebo.
  Interventions: Drug: DFA-02
- DFA-02 placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DFA-02 — Modified release product containing gentamicin and vancomycin for application at the conclusion of surgery after closure of the fascia and prior to skin closure
  Arms: DFA-02
Drug: Placebo — DFA-02 placebo
  Arms: DFA-02 placebo

SUMMARY:
This is a randomized, double-blind, placebo controlled, safety, tolerability, and pharmacokinetic dose escalation Phase II study of DFA-02 in patients undergoing colorectal surgery to evaluate the safety, tolerability and pharmacokinetics of DFA-02.

DETAILED DESCRIPTION:
Despite antibiotic prophylaxis and improvements in surgical techniques, surgical site infections (SSI) still occur. DFA-02 is a novel bioresorbable modified release gel containing both gentamicin and vancomycin to be applied during surgical incision closure for the prevention of surgical site infections (SSIs) in patients undergoing colorectal surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females 18 years of age or older;
2. If female, the patient must be:

   * postmenopausal (if amenorrheic for < 1 year, postmenopausal status must be confirmed by an elevated follicle stimulating hormone [FSH] level > 30 mIU/mL; if amenorrheic for > 1 year, FSH level not required);
   * surgically sterilized (does not have a uterus or has had bilateral tubal ligation); or
   * if of child-bearing potential, she must have a negative serum pregnancy test on entry in the study, and agree to use adequate birth control during the study and for 30 days after the administration of study agent. Medically acceptable contraceptives include: (1) surgical sterilization (such as a tubal ligation or hysterectomy), (2) approved hormonal contraceptives (such as birth control pills, patches, implants or injections), (3) barrier methods (such as a condom or diaphragm) used with a spermicide, or (4) an intrauterine device (IUD);
3. BMI 25-40, inclusive;
4. Scheduled to undergo nonemergent colorectal surgery involving a laparotomy incision of 7 cm or greater (hand-assisted laparoscopic surgery is allowed). List of eligible procedures: left, right or transverse colectomy, segmental/sleeve left colon resection, total abdominal colectomy with ileorectal anastomosis, total abdominal colectomy with ileostomy, total abdominal proctocolectomy, low anterior resection, sigmoid resection, non-emergent Hartmann's procedure, colotomy with polypectomy distal to hepatic flexure, colostomy takedown through laparotomy (not peristomal) incision, ileo-pouch anal anastomosis, abdominal perineal resection of the rectum;
5. Willing and able to give informed consent;
6. Available for evaluation from baseline until final evaluation at 30 days post surgery.

Exclusion Criteria:

1. Known history of hypersensitivity to gentamicin or vancomycin, other aminoglycoside antibiotics or the excipients of the study products (soy bean products or sesame oil);
2. Emergency surgery (urgent surgery is allowed if informed consent is obtained and the study procedures can be performed);
3. Significant concomitant surgical procedure (Note: concomitant appendectomy, cholecystectomy, oophorectomy, and liver biopsy/wedge resection are allowed);
4. Prior laparotomy within the last 60 days of this planned procedure;
5. Planned second laparotomy or colorectal surgical procedure (e.g. colostomy or ileostomy takedown) within 30 days of this planned first procedure;
6. Expectation that a surgical drain will be placed;
7. Preoperative sepsis, severe sepsis, or septic shock;
8. Abdominal wall infection/surgical site infection from previous laparotomy/laparoscopy or for any reason;
9. Active systemic infection or systemic (oral or intravenous) antibiotic therapy within the 1 week prior to the date of surgery other than specified preoperative antimicrobial prophylaxis (Note: single dose antibiotic therapy for dental or other minor procedures is allowed as is the use of oral non-absorbable antibiotics for preoperative bowel decontamination);
10. Requirement for gentamicin or vancomycin preoperative antimicrobial prophylaxis (Note: systemic antibiotic therapy within 72 hours after surgery with gentamicin or vancomycin must be avoided and any systemic antibiotic therapy during that time should be discussed with the Coordinating Center PI or Medical Monitor);
11. Requirement for concomitant use or use during the 30 days prior to Day 1 of any prescription or OTC drug that would interfere with the study or place the patient at undue risk. Concurrent systemic or topical use of other potentially neurotoxic, nephrotoxic, and/or ototoxic drugs, such as gentamicin, cisplatin, cephaloridine, kanamycin, amikacin, polymyxin B, colistin, paromomycin, streptomycin, tobramycin, vancomycin, ethacrynic acid, furosemide, and viomycin, should be avoided;
12. Preoperative evaluation suggests an intra-abdominal process that might preclude full closure of the skin;
13. Ongoing treatment (e.g. chemotherapy, radiation) for non-colorectal cancer;
14. History of significant drug or alcohol abuse within the past year;
15. Serum Creatinine > 1.3 mg/dL
16. Serum Bilirubin > 2.5 times upper limit of normal;
17. History of uncontrolled diabetes mellitus (controlled diabetic patients whose hemoglobin A1c is ≤ 9.0% may be included);
18. Patients who are immunocompromised including but not limited to systemic corticosteroid use or chemotherapy/radiation during the 30 days prior to surgery, organ transplantation, or HIV infection (Note: inhaled corticosteroids are not exclusionary and single dose use of corticosteroids to prevent PONV is allowed.);
19. Any clinically meaningful hearing loss (from Medical History);
20. Clinically exclusionary results on clinical laboratory, ECG, or physical examination including but not limited to positive hepatitis B or C or HIV;
21. Pregnant or lactating, or if of childbearing potential not practicing a birth control method with a high degree of reliability;
22. Refusal to accept medically indicated blood products;
23. Participation within 30 days before the start of this study in any experimental drug or device study, or currently participating in a study in which the administration of investigational drug or device within 60 days is anticipated;
24. Patients with anterior abdominal wall mesh that is not planned to be completely removed during the planned procedure;
25. Unable to participate in the study for any reason in the opinion of the Principal Investigator;
26. Postsurgical life expectancy of less than 30 days, in the Investigator's or Sponsor's opinion;
27. Expected discharge from the hospital less than 3 days after surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-02; Primary Completion 2013-04 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kent Allenby, MD, Study Director — Dr. Reddy's Laboratories
Locations (5):
- United States (5):
  - Florence, Alabama
  - Tampa, Florida
  - Columbus, Ohio
  - Bellaire, Texas
  - Temple, Texas

REFERENCES:
- [Derived] Bennett-Guerrero E, Minkowitz HS, Segura-Vasi AM, Marcet JE, White JA, Corey GR, Allenby KS. A randomized, double-blind, placebo controlled safety, tolerability, and pharmacokinetic dose escalation study of a gentamicin vancomycin gel in patients undergoing colorectal surgery. Perioper Med (Lond). 2016 Jun 16;5:17. doi: 10.1186/s13741-016-0043-2. eCollection 2016. PMID 27313846

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study Period: February 12, 2012 to June 27, 2013. Patients were enrolled at four hospital based sites in the US (Tampa, FL; Temple, Tx; Florence, AL; Houston, TX).
Groups:
- DFA-02: Progressive cohorts of 8 subjects per cohort receiving up to 10, 20 or 30 mL of DFA-02
  DFA-02: Modified release product containing gentamicin and vancomycin for application at the conclusion of surgery after closure of the fascia and prior to skin closure
- DFA-02 Placebo: Progressive cohorts of 2 patients per cohort receiving up to 10, 20 or 30 mL of DFA-02 placebo
Period: Overall Study
Arm/Group | DFA-02 | DFA-02 Placebo
Started | 24 | 6
Completed | 24 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- DFA-02: Progressive cohorts of 8 subjects per cohort receiving up to 10, 20 or 30 mL of DFA-02
- DFA-02 Placebo: Progressive cohorts of 2 subjects per cohort receiving up to 10, 20 or 30 mL of DFA-02 placebo
- Total: Total of all reporting groups
Arm/Group | DFA-02 | DFA-02 Placebo | Total
Number analyzed (Participants) | 24 | 6 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.8 (14.91) | 58.5 (16.7) | 62.0 (15.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 4 | 18
  Male | 10 | 2 | 12
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 21 | 5 | 26
  Black/African American | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 24 | 6 | 30
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 29.8 (4.00) | 27.8 (2.47) | 29.4 (3.79)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Adverse Events, Laboratory, Physical Examination Changes
Description: Safety and tolerability measured by number of patients with adverse events or changes in laboratory or physical examination findings from baseline (DFA-02 application during surgery on Day 1) to 30 days after surgery.
Time Frame: Baseline up to Day 30
Population: As Treated
Measure: Number; unit: Participants
Groups:
- DFA-02: Progressive cohorts of 8 subjects receiving up to 10, 20 or 30 mL of DFA-02
- DFA-02 Placebo: Progressive cohorts of 2 subjects receiving 10, 20 or 30 mL of DFA-02 placebo
Arm/Group | DFA-02 | DFA-02 Placebo
Number analyzed (Participants) | 24 | 6
Participants
  Any Adverse Event | 23 | 6
  Any Serious Adverse Event | 5 | 2
  Related Adverse Event | 3 | 0
  Death | 0 | 1

2. Primary Outcome: Area Under Curve (AUC)
Description: Area under the curve (AUC) of plasma gentamicin and vancomycin levels using sparse sampling from baseline (DFA-02 application during surgery on Day 1) to 4 days after surgery
Time Frame: 1, 6, 24, 48 96 hours post-dose
Population: All Subjects Receiving Active Drug
Measure: Mean (Standard Deviation); unit: mcg/h/mL
Arm/Group | DFA-02 | DFA-02 Placebo
Number analyzed (Participants) | 24 | 0
mcg/h/mL
  Gentamicin AUC (0-t) | 14.2 (12.6) |
  Vancomycin AUC (0-t) | 6.47 (8.12) |

3. Secondary Outcome: Maximal Plasma Concentration (Cmax)
Description: Maximal plasma concentration (Cmax)of gentamicin and vancomycin using sparse sampling from baseline (DFA-02 application during surgery on Day 1) to 4 days after surgery
Time Frame: 1, 6, 24, 48, 96 hours post-dose
Population: All subjects receiving DFA-02 active gel
Measure: Mean (Standard Deviation); unit: mcg/mL
Groups:
- DFA-02: Progressive cohorts of 18 subjects receiving up to 10, 20 or 30 mL of DFA-02
- DFA-02 Placebo: Progressive cohorts of 2 subjects per cohort receiving up to 10, 20 and 30 mL of DFA-02 placebo
Arm/Group | DFA-02 | DFA-02 Placebo
Number analyzed (Participants) | 24 | 0
mcg/mL
  Gentamicin Cmax | 0.642 (0.524) |
  Vancomycin Cmax | 0.164 (0.150) |

4. Secondary Outcome: Renal Function
Description: Changes in serum creatinine from surgery on Day 1 until 14 days after surgery
Time Frame: Baseline up to Day 14
Population: As treated
Measure: Number; unit: Participants
Groups:
- DFA-02: Progressive cohorts of 8 subjects per cohort receiving up to 10, 20 or 30 mL DFA-02
- DFA-02 Placebo: Progressive cohorts of 2 subjects per cohort receiving 10, 20 or 30 mL DFA-02 placebo
Arm/Group | DFA-02 | DFA-02 Placebo
Number analyzed (Participants) | 24 | 6
Participants
  Moderate Elevated Serum Creatinine Day 5 or Day 14 | 1 | 0
  Severe/LifeThreatening Elevated Serum Creatinine | 0 | 0

5. Secondary Outcome: Antibiotic Resistance
Description: Methicillin-resistant Staphylococcus aureus and vancomycin-resistant enterococcus presence at surgery on Day 1 and 5 days after surgery
Time Frame: Baseline up to Day 5
Population: As Treated
Measure: Number; unit: Participants
Groups:
- DFA-02 Placebo: Progressive cohorts of 2 subject per cohort receiving up to 10, 20 or 30 mL DFA-02 placebo
Arm/Group | DFA-02 | DFA-02 Placebo
Number analyzed (Participants) | 24 | 6
Participants
  Nasal MRSA Conversion | 1 | 0
  Rectal Vancomycin Resistant Enterococcus Conversio | 0 | 1

6. Secondary Outcome: Incidence of Surgical Site Infection
Description: The incidence of probable or definite surgical site infection as determined by the Investigator.
Time Frame: Up to 30 Days After Surgery
Population: As treated
Measure: Number; unit: Participants
Groups:
- DFA-02: Progressive cohorts of 8 subjects receiving up to 10, 20 or 30 mL DFA-02
- DFA-02 Placebo: Progressive cohorts of 2 subjects per cohort receiving up to 10, 20 or 30 mL DFA-02 placebo
Arm/Group | DFA-02 | DFA-02 Placebo
Number analyzed (Participants) | 24 | 6
Participants | 6 | 1

ADVERSE EVENTS:
Time Frame: From Informed Consent to 30 Days After Surgery
Arm/Group | DFA-02 | DFA-02 Placebo
Serious Adverse Events (participants affected / at risk) | 5/24 | 2/6
Other Adverse Events (participants affected / at risk) | 23/24 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DFA-02 (N=24) | DFA-02 Placebo (N=6)
Bowel Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anastomotic Leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Small Bowel Anastomotic Leak with Secondary Sepsis
Surgical Site Infection (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Post-operative Bleeding (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Mesenteric Vessel Bleeding
Anastomotic Dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Death (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Anastomotic leak followed by venous thrombosis followed by death
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DFA-02 (N=24) | DFA-02 Placebo (N=6)
Blood and Lymphatic System Disorders (Blood and lymphatic system disorders) | 8 (8) | 2 (2)
Cardiac Disorders (Cardiac disorders) | 9 (9) | 2 (2)
Gastrointestinal Disorders (Gastrointestinal disorders) | 21 (21) | 5 (5)
General Disorders and Administration Site Conditions (General disorders) | 4 (4) | 1 (1)
Hepatobiliary Disorders (Hepatobiliary disorders) | 1 (1) | 0 (0)
Infections and Infestations (Infections and infestations) | 10 (10) | 1 (1)
Injury, Poisoning and Procedural Complications (Injury, poisoning and procedural complications) | 9 (9) | 2 (2)
Investigations (Investigations) | 12 (12) | 3 (3)
Metabolism and Nutritional Disorders (Metabolism and nutrition disorders) | 11 (11) | 2 (2)
Musculoskeletal and Connective Tissue Disorders (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Nervous System Disorders (Nervous system disorders) | 3 (3) | 1 (1)
Psychiatric Disorders (Psychiatric disorders) | 5 (5) | 0 (0)
Renal and Urinary Disorders (Renal and urinary disorders) | 4 (4) | 1 (1)
Respiratory, Thoracic and Mediastinal Disorders (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1)
Skin and Subcutaneous Disorders (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Vascular Disorders (Vascular disorders) | 13 (13) | 2 (2)

LIMITATIONS AND CAVEATS:
Protocol specified cohorts of 10, 20, 30 or 40 mL to be placed after closure of the fascia and prior to skin closure. Experience with 20 and 30 mL dose levels showed that even largest patients would not accommodate 40 mL so that arm was not done.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less